CLINICAL TRIAL: NCT05155553
Title: An Observational Clinical Performance Evaluation Study Testing Residual Specimens of Cerebrospinal Fluid Obtained by Lumbar Puncture From Meningitis/Encephalitis Subjects Using the QIAstat-Dx® Meningitis/Encephalitis Panel
Brief Title: QIAstat-Dx® Meningitis/Encephalitis Panel Performance Evaluation Study
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SMF-DHF-18-0489-002
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Meningitis/Encephalitis
MeSH Terms: conditions — Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — residual specimens of CSF obtained by lumbar puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: QIAstat-Dx® Meningitis/Encephalitis (ME) Panel — The performance of QIAstat-Dx® Meningitis/Encephalitis Panel will be evaluated in comparison with another validated comparator method, followed by bidirectional sequencing using residual specimens of cerebrospinal fluid (CSF) obtained by lumbar puncture from subjects with signs and symptoms of meningitis and/or encephalitis.

SUMMARY:
Study for performance evaluation of the QIAstat-Dx® Meningitis/Encephalitis Panel in comparison with other chosen comparator methods.

DETAILED DESCRIPTION:
This multicenter study aims to evaluate the performance of QIAstat-Dx Meningitis/Encephalitis (ME) Panel with another validated comparator method.

ELIGIBILITY:
Inclusion Criteria:

* Residual specimens (minimum 500μL) of CSF obtained by lumbar puncture from subjects with signs and symptoms of meningitis and/or encephalitis following completion of routine testing Specimen that have not undergone more than 3 freeze/thaw cycles.

Exclusion Criteria:

* Specimens not fitting criteria outlined above.
* CSF obtained from an external ventricular drain or shunt source.
* Lack of clear subject identification or label on residual banked CSF specimen.
* Specimen has been centrifuged.
* Obvious physical damage of banked residual specimen.
* Repeat specimens from the same subject.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects (adults and children) with signs and symptoms of meningitis and/or encephalitis
Sampling Method: Probability Sample
Enrollment: 1524 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
PPA | 6 months
  positive percentage agreement
NPA | 6 months
  negative percentage agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — QIAGEN Gaithersburg, Inc
Locations (1):
- Qiagen, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
all samples are residual and anonymized